CLINICAL TRIAL: NCT00858806
Title: Phase II Explorative Study of Intermittent Imatinib (IM) Treatment (INTERIM) in Elderly Patients With Ph+ Chronic Myeloid Leukemia (CML) Who Achieved a Stable Complete Cytogenetic Response (CCgR) With Standard IM Therapy
Brief Title: Intermittent Imatinib Treatment in Chronic Myeloid Leukemia and Philadelphia Chromosome (Ph+CML) Patients Who Achieved a Complete Cytogenetic Response (CCgR) on Standard Imatinib Therapy
Acronym: INTERIM0407
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Domenico Russo, Full Professor of Hematology, Università degli Studi di Brescia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-005102-42
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intermittent Imatinib (Experimental): Imatinib will be given with the following schedule:
  * 1 week on / 1 week off for the 1st month(weeks 1-4)
  * 2 weeks on / 2 weeks off for the 2nd and the 3rd month (weeks 5-12)
  * 1 month on / 1 month off from the 4th month thereafter (weeks 13 on)
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Imatinib — Intermittent Imatinib administration.
  * 1 week on / 1 week off for the 1st month(weeks 1-4)
  * 2 weeks on / 2 weeks off for the 2nd and the 3rd month (weeks 5-12)
  * 1 month on / 1 month off from the 4th month thereafter (weeks 13 on)
  Other Names: glivec

SUMMARY:
Standard therapy with Imatinib (IM) significantly prolongs the survival of Ph+CML patients who obtain a complete cytogenetic response (CCgR). Elderly patients (i.e., at least 65 years) have similar cytogenetic responses and survival, but they usually show a low compliance. The aim of the study is to evaluate the percentage of elderly patients who maintain a CCgR with intermittent imatinib therapy with respect to standard daily administration.

DETAILED DESCRIPTION:
Objective: The aim of the study is to investigate if the complete cytogenetic response (CCgR) that has been achieved with standard (daily administration) Imatinib (IM) therapy can be maintained with the same dose of IM given intermittently (INTERIM). For the purposes of this study, the term "standard IM therapy" means the daily administration of IM at any dose between 300 and 800mg, whereas, "intermittent IM treatment" (INTERIM), is defined as the same daily dose of IM given one month on/one month off .

The primary objective of the study is to evaluate the proportion of patients who remain in CCgR with INTERIM given for one year.

Study design: This study is an open-label, multicenter, Phase II study of INTERIM for the maintenance of CCgR.

Study Population: Elderly patients (at least 65 years) with Ph+ CML and with stable CCgR after at least 2 years of standard (daily administration ) IM therapy

Treatment Plan STUDY DRUG: Imatinib is registered as Glivec by Novartis Pharma Italy for treatment of patients with Ph+ CML in any phase (CP and AP/BP).

DOSE AND SCHEDULE: Imatinib (Glivec) is given at the same daily dose that was given at the time of the enrollment by the following intermittent schedule:

* 1 week on / 1 week off for the 1st month(weeks 1-4)
* 2 weeks on / 2 weeks off for the 2nd and the 3rd month(weeks 5-12)
* 1 month on / 1 month off from the 4th month thereafter(weeks 13 on)

TREATMENT DURATION: The study has a duration of 12 months. After 12 months of intermittent dose of IM (INTERIM) the patients who are in continuous CCgR are advised to continue study treatment dose (INTERIM) but can go back to pre-study daily dose. Follow up is required indefinitely for all patients.

Efficacy The primary efficacy variable of intermittent dose of IM (INTERIM) is measured by the proportion of patients who maintain a stable CCgR over the whole study period (12 months). For the purposes of this study the monitoring of the cytogenetic response (CgR) status will be evaluated by Fluorescence-in-situ-Hybridization (FISH) of interphase peripheral blood cells (molecular cytogenetic analysis)

OFF TREATMENT EVENTS

Patients go off the study in case of failure:

* Loss of CCgR
* Loss of CHR
* Progression to AP/BP or in case of:
* Patient's refusal
* Documentation of serious adverse events (SAE)
* Protocol violation

OFF-TREATMENT THERAPEUTIC RECOMMENDATIONS

* In case of Loss of CCgR

  * intermittent dose of IM (INTERIM) has to be STOPPED
  * evaluation of additional cytogenetic abnormalities (ACA) by conventional (morphologic) cytogenetics has to be performed
  * mutational analysis of BCR-ABL transcript has to be checked
  * and pre-study IM standard therapy (daily dose administration) has to be RESUMED
* In case of Loss of CHR or Disease Progression to AP/BP

  * intermittent dose of IM (INTERIM) has to be STOPPED
  * and it is recommended to move to investigational available treatments, based on cytogenetic and molecular data
* In case of SAE: it is recommended to discontinue IM forever
* In case of Refusal or Protocol Violation: it is recommended to go back to pre-study IM dose

Concomitant Treatments All patients who are enrolled in this study have already been treated with IM for a minimum of 2 years. Therefore, it is expected that the problems concerning concomitant treatments have already been considered and that the investigators and the patients are familiar with them. However, it is wise to remind that IM is a competitive inhibitor of CYP2D6 and CYP3A4/5. Interactions are possible when IM is administered with drugs whose metabolism is dependent on or which a1ter levels of these P450 cytochrome isoenzymes. When drugs classified as 'substrates' are co-administered with IM, there is the potential for higher concentrations of the 'substrate'. When IM is co-administered with compounds classified as 'inhibitors', increased plasma concentrations of Imatinib is the potential outcome. Particular attention is drawn to the potential interaction between IM and acetaminophen, anticoagulants (especially warfarin) and anticonvulsants.

Visit Schedule, Assessments and Follow-up

* Clinical evaluation and physical examination, including height, weight, vital signs and other relevant findings will be assessed at the time of enrollment (baseline) and every 3 months during the study (12 months).
* Cardiac function assessment will be performed by echocardiography at baseline, and at the end of the study.
* Blood count including Hb, Plt count, WBC and differential will be performed at baseline and will be monitored every 3 months during the study.
* Serum chemistry, including BUN, creatinine, AST, ALT, ALP, bilirubin, Ca, P, K and Mg, total protein concentration and electrophoretic profile, IgG, IgA, IgM concentration will be performed at baseline and every 3 months during the study.
* The cytogenetic response (CgR) status has to be evaluated at baseline and every 3 months during the study

  * At baseline (BL) the cytogenetic response (CgR) status must be evaluated by conventional (morphologic) AND by molecular cytogenetics (FISH) analysis.
  * The monitoring of the cytogenetic response (CgR) status (months 3, 6, 9 and 12) will be evaluated only by Fluorescence-in-situ-Hybridization (FISH) of interphase peripheral blood cells (see section 11.1 page 19). FISH has the potential advantage of i) evaluating many more cells and of using peripheral blood instead of marrow, ii) reducing missing information by conventional morphologic evaluation of marrow cells metaphases, iii) improving the compliance of patients for cytogenetic monitoring.
  * If FISH documents a variation of the baseline value of more than 1%, check again the CgR by a second FISH analysis after 1 months
  * If the second FISH analysis confirms a variation of the baseline value of more than 1%, conventional cytogenetics by evaluation of marrow cells metaphases has to be performed to confirm the Cytogenetic Response Loss (CgR loss) and to check for additional cytogenetic abnormalities (ACA)
* Quantitative molecular assessment of BCR-ABL transcript by RQ-PCR on peripheral blood sample is due at baseline and every 3 months during the study.
* Mutational analysis has to be performed in case of loss of CCgR on marrow cells.
* Follow up is required indefinitely for all patients by standard hematologic, cytogenetic and molecular criteria.

Sample Size This study has been designed according to the optimal Simon's two stage procedure, based on data of the annual rates of treatment failure reported in 454 patients receiving IM in the multicenter, open-label, phase III randomized international study IRIS. The optimal two-stage design to test the null hypothesis that P<= 0.850 versus the alternative that P>= 0.950 has an expected sample size of 33.7 and a probability of early termination of 0.602. If the INTERIM regimen is not effective (in the sense of maintaining a complete cytogenetic response less than 0.85), there is a 0.049 probability of concluding that it is (the target for this value was 0.050). If the INTERIM regimen is effective (in the sense of maintaining a complete cytogenetic response more than 0.85), there is a 0.200 probability of concluding that it is not (the target of this value was 0.200). A total of 78 patients have to be enrolled, 13 in the first stage and 65 in the second stage. The Trial Advisory Committee (TAC) will monitor the accrual and the cytogenetic response status every 3 months and will stop the study if the loss of the CCgR is more than 15.4% and 9.2% in the first and second stage, respectively.

Trial Time Trial time is 12 months. Thereafter, all patients are followed by standard hematologic, cytogenetic and molecular criteria, indefinitely.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed diagnosis of Ph+ CML in CP
2. Age ≥ 65 years old
3. Stable CCgR after at least 2 years of treatment with standard (daily administration) IM therapy documented by 2 consecutive cytogenetic analysis over the last 12 month
4. Karnofsky performance status >50%
5. Written informed consent prior to any study procedures being performed.

Exclusion Criteria:

1. Patients with Ph+ CML in accelerated/blastic phase (AP/BP), or in late CP, previously treated (i.e. IFN alpha+/- low dose Ara-C, Hydroxyurea, allogeneic stem cell transplantation, etc etc.)
2. Age < 65 years old
3. No stable CCgR after at least 2 years of treatment with standard (daily administration) IM therapy documented by 2 consecutive cytogenetic analysis over the last 12 month
4. Karnofsky performance status <50%
5. No written informed consent prior to any study procedures being performed.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 78 (Actual)
Dates: Start 2008-04; Primary Completion 2010-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who remain in CCgR with INTERIM given for one year. | 1 year

SECONDARY OUTCOMES:
Variation of BCR-ABL transcript level | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Prof Domenico Russo, MD, Principal Investigator — Chair of Haematology, Brescia University
Locations (1):
- Chair of Haematology, Bone Marrow Transplant Unit, Brescia, Brescia, Italy

REFERENCES:
- [Derived] Russo D, Martinelli G, Malagola M, Skert C, Soverini S, Iacobucci I, De Vivo A, Testoni N, Castagnetti F, Gugliotta G, Turri D, Bergamaschi M, Pregno P, Pungolino E, Stagno F, Breccia M, Martino B, Intermesoli T, Fava C, Abruzzese E, Tiribelli M, Bigazzi C, Cesana BM, Rosti G, Baccarani M. Effects and outcome of a policy of intermittent imatinib treatment in elderly patients with chronic myeloid leukemia. Blood. 2013 Jun 27;121(26):5138-44. doi: 10.1182/blood-2013-01-480194. Epub 2013 May 15. PMID 23678005